CLINICAL TRIAL: NCT00092729
Title: A Randomized, Placebo-and Active-Comparator-Controlled Study of Etoricoxib 120 mg in the Treatment of Primary Dysmenorrhea
Brief Title: An Investigational Drug Study in the Treatment of Primary Dysmenorrhea (0663-064)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0663-064; MK0663-064; 2004_053
Record Dates: First submitted 2004-09-23; First posted 2004-09-28 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Etoricoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): etoricoxib
  Interventions: Drug: etoricoxib (MK0663)
- 2 (Placebo Comparator): Placebo to match etoricoxib
  Interventions: Drug: Comparator: placebo (unspecified)
- 3 (Active Comparator): naproxen sodium
  Interventions: Drug: Comparator: naproxen sodium

INTERVENTIONS:
Drug: etoricoxib (MK0663) — Two etoricoxib 60 mg tablets and one naproxen sodium 550 mg placebo tablet, single-dose, following onset of moderate-to-severe pain due to primary dysmenorrhea
  Other Names: MK0663
  Arms: 1
Drug: Comparator: placebo (unspecified) — Two etoricoxib 60 mg placebo tablets and one naproxen sodium 550 mg placebo tablet, single-dose, following onset of moderate-to-severe pain due to primary dysmenorrhea
  Arms: 2
Drug: Comparator: naproxen sodium — Two etoricoxib 60 mg placebo tablets and one naproxen sodium 550 mg tablet, single-dose, following onset of moderate-to-severe pain due to primary dysmenorrhea
  Other Names: naproxen sodium
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the pain relieving effect and safety of an investigational drug in women with moderate to severe primary dysmenorrhea (painful menstruation).

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years of age or older suffering from painful menstruation

Exclusion Criteria:

* Women taking medications that are not allowed in the study (such as pain medications, antidepressants, tranquilizers, hypnotics, sedatives, or oral contraceptives).
* Women who are pregnant, breast-feeding or within 6 weeks of giving birth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2002-06-07 (Actual); Primary Completion 2002-12-06 (Actual); Study Completion 2002-12-06 (Actual)

PRIMARY OUTCOMES:
Overall analgesic effect as measured by the total pain relief score over 8 hours post dose (TOPAR8), sum of pain intensity difference over 8 hours post dose (SPID8), and patient's global evaluation at 8 and 24 hours post dose compared with placebo | Up to 8 hours postdose and at 8 and 24 hours postdose, following onset of moderate-to-severe pain due to primary dysmenorrhea for each of three consecutive menstrual cycles
Time to onset, peak, and duration of the analgesic effect compared with placebo | to 24 hours following onset of moderate-to-severe pain due to primary dysmenorrhea for each of three consecutive menstrual cycles

SECONDARY OUTCOMES:
Overall analgesic effect, time to onset, peak, and duration of analgesic effect compared with naproxen sodium | Up to 24 hours following onset of moderate-to-severe pain due to primary dysmenorrhea for each of three consecutive menstrual cycles
Overall analgesic effect, time to onset, peak, and duration of analgesic effect of naproxen sodium compared with placebo | Up to 24 hours following onset of moderate-to-severe pain due to primary dysmenorrhea for each of three consecutive menstrual cycles
Safety and tolerability of etoricoxib as assessed by the number of patients with clinical or laboratory adverse experiences | From randomization through 14 days following the last dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC